CLINICAL TRIAL: NCT04966273
Title: A Prospective, Multi-Center, Non-randomized, Single Arm, Open Label, Study to Evaluate the Safety and Effectiveness of the Biosensors Microcatheter in Coronary Chronic Total Occlusions (CTO) - BIOMICS
Brief Title: Study to Evaluate the Safety and Effectiveness of the Biosensors Microcatheter in Coronary Chronic Total Occlusions (CTO) - BIOMICS
Acronym: BIOMICS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biosensors Europe SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-EU-01
Record Dates: First submitted 2021-06-30; First posted 2021-07-19 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Ischemic Heart Disease
Keywords: Chronic Total Occlusion (CTO); Microcatheter; CTO-PCI
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biosensors Microcatheter (BM) (Experimental): Use of Biosensors Microcatheter
  Interventions: Device: Microcatheter

INTERVENTIONS:
Device: Microcatheter — Only to be used if Biosensor Microcatheter does not perform accordingly
  Other Names: Standard hospital Microcatheter

SUMMARY:
Biosensors, the Sponsor would like to determine if the Biosensors Microcatheter is safe and effective in treating patients with CTO by assessing a composite of in-hospital cardiac death or myocardial infarction and device success (defined as successfully facilitate placement of a guidewire beyond the occluded coronary segment), respectively.

DETAILED DESCRIPTION:
Prospective, multi-center, open-label single-arm trial designed to enroll 100 patients undergoing attempted CTO-PCI at up to 10 centers in the United Kingdom and N. Ireland. For assessment of efficacy, the ability of the BM to successfully facilitate placement of a guidewire beyond the occluded coronary segment will be assessed. Patients will be followed up until hospital discharge or 7 days post index procedure, whichever comes first. For the assessment of safety, the incidence of in-hospital cardiac death or myocardial infarction will be assessed at hospital discharge or 7 days post index procedure, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

1. Adult aged > 18 years
2. Patient understands and has signed the consent form.
3. Patient has an angiographically documented chronic total occlusion (i.e. estimated to be >3 months duration) showing distal TIMI 0 flow. Occlusion with absence of antegrade flow through the lesion and with a presumed or documented duration of 3 months.
4. Suitable candidate for non-emergent PCI
5. Left ventricle ejection fraction > 25%

Exclusion Criteria:

1. Patient unable to give informed consent.
2. Current participation in another study with any investigational drug or device.
3. Known or suspected contrast allergy.
4. in-stent CTO.
5. Planned treatment of a second CTO during the index procedure
6. Intolerance to Aspirin and/or inability to tolerate a second antiplatelet agent (Clopidogrel or Prasugrel or Ticagrelor).
7. Recent major cerebrovascular event (history of stroke or TIA within 1 month)
8. Renal insufficiency (serum creatinine of > 200μmol/L)
9. Active gastrointestinal bleeding
10. Active infection or fever that may be due to infection
11. Life expectancy < 2 years due to other illnesses
12. Significant anaemia (haemoglobin < 10.0g/L)
13. Severe uncontrolled systemic hypertension (> 240 mmHg within 1 month of procedure)
14. Severe electrolyte imbalance
15. Congestive heart failure [New York Heart Association (NYHA) Class III\IV] CSA Class IV.
16. Unstable angina requiring emergent PCI or coronary artery bypass graft (CABG)
17. Recent myocardial infarction (MI) (within the past one week)
18. Unwillingness or inability to comply with any protocol requirements
19. Subject is pregnant or nursing. Female subjects of child-bearing potential must have a negative pregnancy test done within 7 days prior to the index procedure per site standard test.
20. Extensive prior dissection from a coronary guidewire use
21. Drug abuse or alcoholism.
22. Patients under custodial care.
23. Bleeding diathesis or coagulation disorder
24. Kawasaki's disease or other vasculitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2022-03-18 (Actual); Primary Completion 2023-01-03 (Actual); Study Completion 2023-01-03 (Actual)

PRIMARY OUTCOMES:
Efficacy: Percentage of patients with device success | Follow-up only up to hospital discharge or 7 days maximum post procedure, whichever comes first.
  Device success defined as successful placement of a guidewire in the vessel across the occluded coronary segment
Safety: Percentage of patients with composite of in-hospital cardiac death or myocardial infarction. | Follow-up only up to hospital discharge or 7 days maximum post procedure, whichever comes first.
  Composite of in-hospital cardiac death or myocardial infarction.

SECONDARY OUTCOMES:
Percentage of patients with technical success | Follow-up only up to hospital discharge or 7 days maximum post procedure, whichever comes first.
  Technical success is defined as achievement of TIMI grade 2 antegrade flow with less than 50% residual stenosis of the target CTO lesion at procedure end
Percentage of patients with procedural success | Follow-up only up to hospital discharge or 7 days maximum post procedure, whichever comes first.
  Procedural success defined as technical success plus the absence of in-hospital MACE (death, myocardial infarction or clinically-driven target vessel revascularization (cd TVR)
Percentage of patients with crossing success | Follow-up only up to hospital discharge or 7 days maximum post procedure, whichever comes first.
  Crossing success defined as the BM crossing the lesion

OTHER OUTCOMES:
Percentage of patients with device-related perforation | Follow-up only up to hospital discharge or 7 days maximum post procedure, whichever comes first.
  Device-related perforation at the site of target coronary lesion and/or its proximal reference segment including donor artery or collateral
Percentage of patients with device failure | Follow-up only up to hospital discharge or 7 days maximum post procedure, whichever comes first.
  Device failure is defined as:
  * any evidence of fracture of any part of the microcatheter,
  * evidence of wire puncture of any part of the device
  * and/or evidence of a fragment being retained in the body of the patient after a procedure.

CONTACTS AND LOCATIONS:
Overall Officials: James Sprattt, Professor, Principal Investigator — St. George's Hospital, London; Margaret MCENTEGART, Dr., Principal Investigator — Golden Jubilee National Hospital
Locations (9):
- United Kingdom (9):
  - Basildon and Thurrock University, Basildon, Essex
  - Golden Jubilee Hospital,, Clydebank, Glasgow, Scotland
  - St George's Hospital, Blackshaw Road,, London, Tooting
  - Royal Victoria Hospital, Belfast
  - Bristol Heart Institute, UHBW NHS Trust, Bristol
  - London North West University Healthcare Nhs Trust, Harrow
  - Leeds General Infirmary, Leeds
  - Glenfield Hospital, Leicester
  - University Hospital of Wales, Wales

IPD SHARING:
Plan to Share IPD: Yes
The emphasis in all scientific publications and presentations will be placed on the endpoint at discharge.